CLINICAL TRIAL: NCT05631782
Title: Effects of Shenkang Decoction on Creatinine and Blood Urea Nitrogen in Chronic Renal Failure Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Effects of Shenkang Decoction on Creatinine and Blood Urea Nitrogen in Chronic Renal Failure Hemodialysis Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First People's Hospital of Zunyi (Other)
Responsible Party: Principal Investigator, Wenfu Cao, Director, The First People's Hospital of Zunyi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Caowenfu590
Record Dates: First submitted 2022-11-10; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Chronic Renal Failure; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): losartan tablets were taken orally (J20180054; Hangzhou Merck Pharmaceutical Co., Ltd.; specification 50 mg) at a dose of 50 mg per day. Furosemide was injected intravenously (TCM approved by H41021056; Suicheng Pharmaceutical Co., Ltd.; specification 20 mg: 2mL) at a dose of 100 mg per day. Uremic clearance granule was mixed with water and taken (Z20073256; Kangchen Pharmaceutical (Khorgos) Co., Ltd.; Specification 5 g) at a dose of 5 g at 6:00,12:00 and 10 g at 22:00 every day. Treatment lasted for 10 - 14 days.
  Interventions: Drug: Shenkang decoction
- Treatment group (Experimental): Shenkang decoction prescription: 15 g of semen cuscutae, herba epimedii and pericarpium arecae. 20 g of Eucommia ulmoides Oliv., radix astragali, codonopsis pilosula, salvia miltiorrhiza, tuckahoe, atractylodes macrocephala, Chinese yam, honeysuckle, polyporus umbellatus and dandelion. 15 g of safflower. 12 g of processed Fuzi. 10 g of Radix phytolaccae and sage. Golden cherry son 20 g and puzzle kernel 15 g were added to patients with frequent proteinuria and nocturia took. Yellow cypress 15 g was added to patients with damp-heat in lower-Jiao. The decoction pieces were purchased from the Traditional Chinese Medicine and Pharmacy Department of the First People's Hospital of Zunyi City. They were decocted by computer automatic decocting machine (model) and divided into 150 mL / bag, taken orally, once in the morning, noon and evening, 3 times / day, 1 bag / time, one pair a day. Treatment lasted for 10 - 14 days.
  Interventions: Drug: Shenkang decoction

INTERVENTIONS:
Drug: Shenkang decoction — Given Shenkang decoction on the basis of the above treatment. Shenkang decoction prescription: 15 g of semen cuscutae, herba epimedii and pericarpium arecae. 20 g of Eucommia ulmoides Oliv., radix astragali, codonopsis pilosula, salvia miltiorrhiza, tuckahoe, atractylodes macrocephala, Chinese yam, honeysuckle, polyporus umbellatus and dandelion. 15 g of safflower. 12 g of processed Fuzi. 10 g of Radix phytolaccae and sage. Golden cherry son 20 g and puzzle kernel 15 g were added to patients with frequent proteinuria and nocturia took. Yellow cypress 15 g was added to patients with damp-heat in lower-Jiao. The decoction pieces were purchased from the Traditional Chinese Medicine and Pharmacy Department of the First People's Hospital of Zunyi City. They were decocted by computer automatic decocting machine (model) and divided into 150 mL / bag, taken orally, once in the morning, noon and evening, 3 times / day, 1 bag / time, one pair a day. Treatment lasted for 10 - 14 days.

SUMMARY:
To explore the clinical effect of Shenkang Decoction in chronic renal failure (CRF) patients with hemodialysis (HD).

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of western medicine meets the diagnostic criteria of chronic kidney failure in Internal Medicine
* the diagnosis of TCM meets the diagnostic criteria of the disease in the Guiding Principles for Clinical Research of New Chinese Medicine.
* The patient is over 18 years old,
* can think independently and have civil conduct,
* strictly follow the doctor's advice,
* maintain stable condition and regular HD treatment.

Exclusion Criteria:

* Patients with HD time of no more than three months, severe uncontrolled infection, other malignant diseases, heart, liver, brain, and digestive system dysfunction, mental diseases such as dementia or depression;
* contraindications to HD or contraindications to the study (Shock or systolic blood pressure below 80mm/Hg, severe bleeding or a tendency to bleed, serious infection such as sepsis, or a blood-borne infection, advanced tumor, extremely debilitating or not cooperating with doctor)
* drug allergy, chronic use of glucocorticoids, and immunosuppressants.
* women during pregnancy or lactation.

Ages: 52 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-26 (Actual)

PRIMARY OUTCOMES:
Renal function index | 8 min
  The AU5800 fully automatic biochemical analyzer produced by Beckman Coulter Co., Ltd. was selected for renal function index determination. peripheral venous blood (3-5 mL) was extracted before and after treatment, and Cre and urea nitrogen were measured after centrifugation
TCM syndrome points | 14 days
  According to the relevant contents of the Clinical Guiding Principles of New Chinese Medicine13, clinical symptoms of shortness of breath, fatigue, anorexia, chills, abdominal fullness and distension, unsolid stool, and weak waist were evaluated.
Nutritional status index | 14days
  In patients, 3 mL of fasting venous blood was collected and given anticoagulant treatment. The total serum protein, serum albumin, hemoglobin, and total red blood cells were measured by Mindray automatic biochemical analyzer (model BS-280, Shenzhen Mindray Bio-Medical Electronics Co., LTD.).
Dialysis adequacy judgment index | 14 days
  The urea dynamic model was used to evaluate the overall urea clearance judgment of a single dialysis effect, and Kt / V was calculated according to the Daugirdas formula. Kt / V= -ln (BUN before dialysis / BUN after dialysis-0.008 t) + (4-3.5 BUN before dialysis /BUN after dialysis) ultrafiltration volume / dialysis body weight. Long-term dialysis components are protein catabolism rate (calculated by Gotch formula) and time-average urea concentration (calculated by Lowrie formula). Protein catabolism rate = 9.35G×0.29Vt.
Treatment efficiency | 14 days
  The efficacy of the two groups was compared with the TCM syndrome points and the biochemical examination indexes.
General physical examination | 14 days
  Including heart rate, blood pressure, breathing, pulse, and urine volume. Urine routine, blood routine, stool routine, liver and kidney function testing, and electrocardiogram monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Zunyi, Zunyi, China